CLINICAL TRIAL: NCT01553188
Title: A Phase II Multicenter Study of AMG 386 and Abiraterone in Metastatic Castration Resistant Prostate Cancer
Brief Title: AMG 386 and Abiraterone for Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120079; 12-C-0079
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Prostatic Neoplasms; Prostate Cancer; Neoplasm, Prostate; Neoplasm,Prostatic
Keywords: Anti-Angiogenesis; Ang 1; Ang 2; Peptide-Fc fusion protein; Small Molecule
MeSH Terms: conditions — Prostatic Neoplasms | interventions — trebananib; abiraterone; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abiraterone, Prednisone and AMG (Experimental): Abiraterone and prednisone will be given with maximum tolerated dose (MTD) of Trebananib (AMG)
  Interventions: Drug: AMG 386; Drug: Abiraterone; Drug: Prednisone
- Abiraterone and Prednisone only (Active Comparator): Abiraterone and prednisone only
  Interventions: Drug: Abiraterone; Drug: Prednisone
- Run in (Other): Dose escalation phase to determine MTD of AMG
  Interventions: Drug: AMG 386; Drug: Abiraterone

INTERVENTIONS:
Drug: AMG 386 — AMG 386 dose will be calculated using the subjects actual body weight (Kg). Supplied in 240 mg v will be administered as an intravenous (IV) infusion using an intravenous infusion pump given over a 60-minute period.
  Other Names: Trebananib
  Arms: Abiraterone, Prednisone and AMG; Run in
Drug: Abiraterone — A 1,000 mg dose of abiraterone should be taken orally once daily
  Other Names: Zytiga
Drug: Prednisone — Prednisone should be taken orally either, at 5mg twice a day for each dose or 10 mg once a day a patients preference.
  Other Names: Deltasone
  Arms: Abiraterone and Prednisone only; Abiraterone, Prednisone and AMG

SUMMARY:
Background:

* Advanced prostate cancer is treated with surgery or drugs that lower the levels of androgens (male hormones) in the body. However, some cancers become resistant to this treatment. These types of cancers are known as castration-resistant prostate cancers.
* Interfering with the growth of blood vessels that feed tumors can slow prostate cancer growth. Trebananib (AMG 386), a new anticancer drug, targets the blood vessels that feed tumors. It has been tested for different types of cancer, but not for prostate cancer. Researchers want to see if AMG 386 can slow disease progression in men with castration-resistant prostate cancer. AMG 386 will be given with abiraterone and prednisone, two drugs that are also used to treat advanced prostate cancer.

Objectives:

- To test the safety and effectiveness of AMG 386 with abiraterone for castration-resistant prostate cancer.

Eligibility:

- Men at least 18 years of age with castration-resistant prostate cancer.

Design:

* Participants will be screened with a physical exam, medical history, and imaging studies. Blood and urine samples will also be collected.
* Participants will be separated into two groups.
* The first group will have AMG 386 once per week for a total of four doses during a 28-day cycle. They will also take abiraterone once a day and prednisone twice a day, every day of the cycle.
* The second group will not have AMG 386. They will take abiraterone once a day and prednisone twice a day, every day of the 28-day cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take the study drugs as long as the disease does not progress and there are no severe side effects.

DETAILED DESCRIPTION:
Background:

* Inhibition of angiogenesis, either as a stand-alone approach or in combination with chemotherapy, has demonstrable antitumor efficacy against castration-resistant prostate cancer (CRPC) and there are several antiangiogenic agents that are now in clinical trials in this population of patients.
* AMG 386 is a novel peptide-Fc fusion protein. The molecule is a non-glycosylated homodimer engineered by fusing an Immunoglobulin gamma-1 heavy chain constant region, partial (IgG1 Fc) domain to 4 copies of an anti-angiopoietin 2 (Ang2) peptide. AMG 386 sequesters Ang1 and Ang2, thereby preventing their interaction with Tie2 and inhibiting tumor endothelial cell (EC) proliferation and tumor growth.
* Abiraterone acetate is a small molecule that irreversibly inhibits Cytochrome P450 17A1 (CYP17), a rate-limiting enzyme in androgen biosynthesis, to block residual androgen synthesis in the adrenal gland and tumor cells.
* Previous studies have demonstrated that in vivo alterations of testosterone levels regulate the expression of vascular endothelial growth factor (VEGF), fibroblast growth factor (FGF), and angiopoietin family members. Dual targeting of the androgen and angiogenic axis represents a novel approach as a potential targeted therapy for patients with metastatic castration-resistant prostate cancer (CRPC).

Objectives:

-To estimate the treatment effect as measured by progression free survival (PFS) in patients treated with AMG 386 plus abiraterone/prednisone relative to abiraterone/prednisone alone.

Eligibility:

-Patients with progressive, metastatic CRPC with radiographic evidence of progression after primary therapy (surgery or radiotherapy) and adequate androgen deprivation therapy.

Design:

* This is an open-label, randomized, phase II multicenter trial with a two-part design and a planned accrual of 88 patients.
* An initial run-in phase of AMG 386 will be conducted with 15mg/kg weekly escalating to 30mg/kg weekly to establish the MTD. The decision on declaration of a safe and tolerable dose during this run-in phase will lead to the second part of the study consisting of a randomized comparison of abiraterone/prednisone plus AMG 386 (at the established maximum tolerated dose (MTD)) vs. abiraterone/prednisone alone.
* AMG 386 will be administered intravenously every week, on days 1, 8, 15 and 22 of each 28-day cycle. Abiraterone acetate will be self-administered once daily by mouth and prednisone will be self-administered by mouth either twice per day at 5 mg per dose or once per day at 10 mg per dose as the patient prefers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have metastatic, progressive, castrate-resistant prostate cancer (CRPC) with radiographic evidence of disease that has continued to progress radiographically or biochemically (rising prostatic specific antigen (PSA) levels on successive measurements) despite adequate androgen-deprivation therapy. If patients had been on flutamide, disease progression is documented 4 weeks or more after withdrawal. For patients on bicalutamide or nilutamide disease progression is documented 6 or more weeks after withdrawal. Flutamide, nilutamide and bicalutamide disease progression requirements only apply to patients who have been on these drugs for at least the prior 6 months.
* Histopathological confirmation of prostate cancer by the Laboratory of Pathology of the National Cancer Institute (NCI) or Walter Reed National Military Medical Center prior to entering this study. Patients enrolled at participating sites may have histopathological confirmation at the enrolling center prior to entering the study. Patients whose pathology specimens are no longer available may be enrolled if the patient has a clinical course that is consistent with prostate cancer and available documentation from an outside pathology laboratory of the diagnosis. All efforts should be made to have the material forwarded to the research team for use in correlative studies in cases where original tissue blocks or archival biopsy material is available.
* Patients must have metastatic disease, defined as at least one lesion on bone scan or at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam.
* Patients participating in the study must have Metastatic Castration-Resistant Prostate Cancer (mCRPC).
* Patients who have received docetaxel plus androgen deprivation therapy (ADT) for metastatic castrate sensitive prostate cancer are eligible for the study. (Patients may enroll as long as they did not have progressive disease while on docetaxel and are 6 months removed from treatment, with all treatment related toxicities resolving to at least grade 1.)
* Patients may not have had more than 7 days of treatment with ketoconazole by mouth in the past 6 months.
* Males greater than or equal to 18 years of age. Because no dosing or adverse event data are currently available on the use AMG 386 in combination with abiraterone in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 for run-in phase; ECOG less than or equal to 1 for randomized phase.
* Life expectancy of > 3 months for the run in phase and > 6 months for the randomized phase.
* Adequate bone marrow, hepatic, and renal function with:

  * Leukocytes greater than or equal to 3000/mu L
  * Absolute neutrophil count (ANC) greater than or equal to 1500/mu L
  * Platelets greater than or equal to 100000/mu L
  * Total bilirubin less than or equal to 1.5 times institutional upper limits of normal
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 times institutional upper limits of normal
  * Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) less than or equal to 1.5 times upper limits of normal (ULN) per institutional laboratory range and international normalized ratio (INR) less than or equal to 5
  * Creatinine less than or equal to 1.5 times institutional upper limits of normal

OR

* Creatinine clearance of >40 mL/min per 24 h urine collection or calculated according to the Cockcroft-Gault formula

  ---Creatinine clearance (CrCl) (mL/min) = (((140-age) times actual body weight (kg))/(72 x serum creatinine (mg/dL)))*(x 0.85 for females)
* Urinary protein less than or equal to 30 mg/dL in urinalysis or less than or equal to1+ on dipstick, unless quantitative protein is <1000 mg in a 24h urine sample

  * Generally well-controlled blood pressure with systolic blood pressure less than or equal to 140 mmHg AND diastolic blood pressure less than or equal to 90 mmHg prior to enrollment. The use of antihypertensive medications to control hypertension is permitted.
  * Must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 Common Terminology Criteria in Adverse Events (CTCAE) version 4 or has returned to baseline. Alopecia >grade 1 is permitted.
  * The effects of AMG 386 on the developing human fetus are unknown. For this reason and because inhibitors of angiogenesis as well as other therapeutic agents used in this trial are known to be teratogenic, men must agree to use adequate contraception

(hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating

physician immediately. Men treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of AMG 386 administration.

-Must have the ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy for metastatic castration-resistant prostate cancer.
* History or presence of known central nervous system metastases.
* History of venous or arterial thromboembolism within 12 months prior to enrollment/randomization.
* History of clinically significant bleeding within 6 months of enrollment/randomization.
* Currently or previously treated with AMG 386, or other molecules that primarily inhibit the angiopoietins or Tie2 receptor.
* Clinically significant cardiovascular disease within 12 months prior to enrollment/randomization, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication or placement of percutaneous transluminal coronary angioplasty/stent.
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery.
* Minor surgical procedures, placement of tunneled central venous access device within 3 days prior to randomization/enrollment.
* Treatment within 30 days prior to enrollment with the following: cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, methotrexate, azathioprine, rapamycin, and targeted immune modulators such as abatacept (CTLA-4-Ig), adalimumab,

alefacept, anakinra, belatacept (LEA29Y), efalizumab, etanercept, infliximab, or rituximab.

* Patients who have had large field radiotherapy must wait 2 weeks prior to entering the study.
* Non-healing wound, ulcer (including gastrointestinal), or fracture.
* Contraindication to steroid use or history of allergic reactions attributable to the study compounds.
* History of allergic reactions to bacterially-produced proteins.
* Previously diagnosed with another malignancy, within the past two years with the exception of non-melanoma skin cancers or non-invasive bladder cancer.
* Patients who have not yet completed at least 28 days (30 days for prior monoclonal antibody therapy) since receiving other investigational drugs.
* Inability to absorb abiraterone after oral administration (i.e., previous major gastrointestinal surgery or gastrointestinal disease resulting in malabsorption).
* Use of ketoconazole, itraconazole, ritonavir, cyclosporine, carbamazepine, phenytoin, phenobarbital within 2 weeks prior to and while on study therapy.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the study agents. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive

therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

* Uncontrolled intercurrent illness or infections, unstable angina pectoris, cardiac arrythmias, renal dysfunction, or psychiatric illness/social situations that would limit compliance with study requirements.
* Have had treatment with docetaxel for the treatment of metastatic castrate-sensitive prostate cancer within 6 months before the first dose of study enrollment.
* Have had progression of prostate cancer on prior docetaxel treatment for castrate sensitive disease.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02-08 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goktas S, Crawford ED. Optimal hormonal therapy for advanced prostatic carcinoma. Semin Oncol. 1999 Apr;26(2):162-73. PMID 10597727
- [Background] Gulley J, Dahut WL. Chemotherapy for prostate cancer: finally an advance! Am J Ther. 2004 Jul-Aug;11(4):288-94. doi: 10.1097/01.mjt.0000133582.68709.e3. PMID 15266221
- [Background] Berthold DR, Sternberg CN, Tannock IF. Management of advanced prostate cancer after first-line chemotherapy. J Clin Oncol. 2005 Nov 10;23(32):8247-52. doi: 10.1200/JCO.2005.03.1435. PMID 16278480
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0079.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An initial run-I phase of AMG 386 will be conducted with 15mg/kg weekly escalating to 30mg/kg weekly to establish the maximum tolerated dose.
Groups:
- DL 1 Run in - 15mg/kg; DL 2 Run in - 30mg/kg: Dose escalation phase to determine MTD of AMG
  AMG 386: AMG 386 dose will be calculated using the subjects actual body weight (Kg).
  Abiraterone: A 1,000 mg dose of abiraterone should be taken orally once daily
  DL 1 AMG is 15 mg/kg DL 2 AMG is 30 mg/kg
  The randomized portion is 30 mg/kg.
Period: Overall Study
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only
Started | 3 | 6 | 16 | 11
Completed | 2 | 5 | 14 | 11
Not Completed | 1 | 1 | 2 | 0
Not completed — Patient choice | 1 | 0 | 0 | 0
Not completed — Intercurrent illness and adverse event | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only | Total
Number analyzed (Participants) | 3 | 6 | 16 | 11 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 2 | 3 | 14
  >=65 years | 0 | 0 | 14 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (1.8) | 62.9 (8.7) | 74.85 (7.44) | 66.05 (9.87) | 69.13 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 6 | 16 | 11 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not meeting definition for Hispanic or Latino | 3 | 6 | 16 | 10 | 35
  Mexican, Puerto Rican, Cuban, Central or So Amer. | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 4 | 5 | 0 | 9
  White | 3 | 2 | 10 | 11 | 26
  Unknown | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 16 | 11 | 36
OnStudy Prostatic Specific Antigen (PSA) [Count of Participants; unit: Participants] — Prostatic Specific Antigen (PSA) reference range is 4.0 ng/mL
  Participants
    >4.0 mg/mL | 3 | 6 | 0 | 0 | 9
    <4.0 mg/mL | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first. Clinical progression is assessed by the Response Criteria in Solid Tumors (RECIST) and is at least a 20% increase in the sum of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Median potential follow-up of 50.3 months
Population: One patient of the 9 (i.e., Run-in in Participant Flow) was not evaluable for responses as we previously defined through the document. Thus, it cannot be included in the PFS assessment. Patient came off the trial early for other reasons.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only
Number analyzed (Participants) | 2 | 6 | 16 | 11
Months | 2.8 [1.9 to 3.6] | 9.0 [1.8 to 29.1] | 11.5 [5.5 to 19.2] | 10.1 [2.7 to 13.7]
Statistical Analysis 1: Comparison: Abiraterone, Prednisone and AMG; Test type: Superiority; p = 0.44, Log rank two-tailed p-value

2. Secondary Outcome: Radiographic Progression Free Survival
Description: Radiographic progression free survival is defined as the duration of time from start of treatment to time of radiographic progression by computed tomography (CT) scan (or magnetic resonance imaging (MRI)) or bone scan. Progression is a minimum of two new lesions observed on bone scan. The minimum size for a measurable lesion on CY and MRI should be twice the slice thickness based on the assumption that CT slice thickness is 500 or less.
Time Frame: Median potential follow-up of 50.3 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only
Number analyzed (Participants) | 2 | 6 | 16 | 11
Months | 2.7 [1.8 to 3.6] | 9.0 [1.8 to NA] — The undefined value is because of the small numbers and the data. It is not estimable. | 13.7 [8.2 to 19.2] | 10.6 [2.7 to 20.1]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is the time between the first day of treatment to the day of death.
Time Frame: Time between the first day of treatment to the day of death, approximately 50.3 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only
Number analyzed (Participants) | 2 | 6 | 16 | 11
Months | 11.1 [5.4 to 16.8] | 27.9 [10.7 to NA] — The undefined value is because of the small numbers and the data. It is not estimable. | 31.1 [18.8 to 43.2] | 25.5 [8.1 to 34.8]
Statistical Analysis 1: Comparison: DL 1 Run in - 15mg/kg vs Abiraterone, Prednisone and AMG; Test type: Superiority; p = 0.26, Log rank two-tailed p-value

4. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 65 months and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only
Number analyzed (Participants) | 3 | 6 | 16 | 11
Participants | 3 | 6 | 16 | 11

5. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is defined as the highest dose studied for which the incidence of dose limiting toxicity was less than 33%.
Time Frame: First 28 days of treatment
Measure: Number; unit: mg/kg
Groups:
- All Participants: All participants who had at least one dose of Abiraterone, prednisone, and/or Trebananib (AMG 386).
Arm/Group | All Participants
Number analyzed (Participants) | 36
mg/kg | 30

6. Other Pre Specified Outcome: Dose Limiting Toxicity (DLT)
Description: DLTs are defined as any grade 3 or higher hematologic (excluding anemia) or non-hematologic toxicity considered to be possible related to AMG 386. Any treatment related adverse events that lead tor reduction of dose exposure of either agent (duration or dose) by >50% in cycle 1 will be considered a DLT.
Time Frame: First 28 days of treatment
Population: Per protocol, only participants in the Run-in phase were evaluated for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 65 months and 7 days.
Arm/Group | DL 1 Run in - 15mg/kg | DL 2 Run in - 30mg/kg | Abiraterone, Prednisone and AMG | Abiraterone and Prednisone Only
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/6 | 4/16 | 3/11
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 14/16 | 11/11
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 16/16 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL 1 Run in - 15mg/kg (N=3) | DL 2 Run in - 30mg/kg (N=6) | Abiraterone, Prednisone and AMG (N=16) | Abiraterone and Prednisone Only (N=11)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 6 (6) | 8 (8)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — disease progression
Confusion (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DL 1 Run in - 15mg/kg (N=3) | DL 2 Run in - 30mg/kg (N=6) | Abiraterone, Prednisone and AMG (N=16) | Abiraterone and Prednisone Only (N=11)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 9 (14) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (6) | 3 (5)
Edema limbs (General disorders) | 0 (0) | 5 (10) | 14 (33) | 7 (12)
Fatigue (General disorders) | 1 (1) | 3 (3) | 8 (14) | 5 (7)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Genital edema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle weakness lower limb (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 3 (5)
Pain (General disorders) | 1 (1) | 2 (2) | 3 (7) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (5) | 3 (8)
Weight gain (Investigations) | 1 (1) | 3 (3) | 11 (28) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (5) | 3 (5)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Edema trunk (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 6 (12) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — subconjunctival hemorrhage s/p fall
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — skin thinning
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 4 (9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (6) | 5 (12)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 4 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 3 (6) | 4 (9)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Nervous system disorders - Other, restless legs (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Skin and subcutaneous tissue disorders - Other, abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 6 (8)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — cerumen removed from auditory canal
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Leg muscle cramps
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Baker's cyst; open neck lesion
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT01553188/Prot_SAP_ICF_000.pdf